CLINICAL TRIAL: NCT04418570
Title: Hormonal and Inflammatory Biomarkers and Response to a Cognitive Remediation Therapy in Recent-onset Psychosis: Randomized, Cross-over, Single-blind, Pilot Clinical Trial
Brief Title: Hormonal and Inflammatory Biomarkers and Response to Cognitive Remediation in Recent-onset Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Javier Labad, Principal investigator, Corporacion Parc Tauli
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PI15/01386
Record Dates: First submitted 2020-05-24; First posted 2020-06-05 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Psychotic Disorders
Keywords: early psychosis; cortisol; inflammation; thyroid; prolactin; cognitive rehabilitation; cognitive remediation
MeSH Terms: conditions — Psychotic Disorders; Inflammation; Thyroid Diseases | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive remediation (Experimental): Computerized cognitive remediation through Neuropersonal Trainer software, 1.5 h per session twice a week for 12 weeks (36 h of total duration).
  Participants will also attend the Early Intervention Service for Psychosis with visits by a psychiatrist, clinical psychologist, social worker, or nurse as scheduled.
  Interventions: Behavioral: cognitive remediation; Other: attendance to an Early Intervention Service for Psychosis
- Treatment as usual (Other): Participants will attend the Early Intervention Service for Psychosis with visits by a psychiatrist, clinical psychologist, social worker, or nurse as scheduled.
  Interventions: Other: attendance to an Early Intervention Service for Psychosis

INTERVENTIONS:
Behavioral: cognitive remediation
  Arms: Cognitive remediation
Other: attendance to an Early Intervention Service for Psychosis

SUMMARY:
This study aims to explore whether hormones or inflammatory markers are associated with cognitive changes following cognitive remediation therapy (CRT) in people with a recent-onset psychotic disorder.

The following biomarkers for treatment response will be considered: hormones related to the hypothalamic-pituitary-adrenal (HPA) axis (plasma cortisol, cortisol awakening response, diurnal cortisol slope, salivary cortisol at assessment), free thyroxine (F-T4), prolactin, or inflammatory markers.

This study was designed as a pilot clinical trial in order to know the feasibility of the intervention and to calculate the effect sizes of different hormonal and inflammatory variables on cognition. This approach would allow the design of future larger clinical trials to test specific hypotheses generated with this study.

DETAILED DESCRIPTION:
Cognitive dysfunction is a core feature of schizophrenia experienced by approximately 75% of the patients. It may occur at the early stages of psychosis, and it is usually unaltered despite positive symptom remission. Cognitive function at psychosis onset is what most strongly predicts worse long-term overall functioning as well as worse functionality in social and occupational areas. Cognitive remediation therapy (CRT) is an intervention targeting cognitive deficit using scientific principles of learning with the ultimate goal of improving functional outcomes. It has been shown to have a significant impact on cognition with medium effect sizes. Some studies have shown improvements in recent-onset psychosis patients reporting moderate to large effects on cognitive outcomes, such as verbal and working memory, visuospatial ability, psychosocial functioning, problem-solving, or executive functioning.

Although CRT is an effective approach, there are data showing that 25-44% of the participants receiving this intervention will not improve. To date, only a limited number of studies have considered potential biomarkers that could predict the treatment response. Hormones and inflammatory markers are potential biomarkers that could moderate the response to CRT because they play important roles in cognitive function in psychiatric and non-psychiatric populations. Previous studies have suggested that hypothalamic-pituitary-adrenal axis hormones (e.g. cortisol), prolactin, thyroid hormones, and inflammatory markers are associated with cognitive performance.

Twenty-eight patients with a recent-onset psychosis aged between 18 and 40 years old and with less than 3 years of duration of the illness will be recruited. Psychotic disorders will include the following DSM-IV diagnosis: schizophrenia, schizoaffective disorder, bipolar disorder, or psychotic disorder not otherwise specified. The patients will be recruited from the Early Intervention Service from Hospital Universitari Parc Taulí Sabadell, (Spain). All participants will be outpatients with stable illness (<4 points in each positive item of the Positive and Negative Syndrome Scale (PANSS) and being on community treatment for at least 4 weeks).

A randomized crossover clinical trial will be performed: one group will first receive computerized CRT (n=14) for three months, and the other group will receive treatment as usual (TAU) in the Early Intervention Service (n=14). Afterward, patients will switch arms to receive alternative intervention.

The intervention will consist of a computerized CRT through Neuropersonal Trainer software (Fernandez-Gonzalo et al. 2015). This includes two rehabilitation modules: 1) the Cognition Module, that addresses the following cognitive domains: on sustained, selective and divided attention; verbal, spatial, visual and working memory; and executive functions including inhibition, sequence and planning; and 2) the Social Cognition Module, which allows working different aspects of emotional processing, the theory of mind and cognitive biases through 43 multimedia-based tasks. Both modules have different levels of complexity. Each CRT session will be individualized to the cognitive needs of each patient by an expert neuropsychologist. The professional can adjust the difficulty level in each treatment session based on the participant baseline cognitive profile and his/her task performance in previous treatment sessions. The neuropsychologist will be guiding the sessions, assuring the understanding of the different tasks, and individually coaching every patient to achieve the correct performance.

A fasting morning blood sample (drawn between 8 a.m. and 10 a.m.) will be obtained for all participants at baseline, at 12 weeks and at 24 weeks of follow-up, for determining cortisol, prolactin, hypothalamic-pituitary-thyroid axis hormones (thyroid-stimulating hormone [TSH] and free thyroxine [F-T4]), and inflammatory markers (IL-6, TNF-alpha, leukocyte count). Saliva samples will be collected for exploring hypothalamic-pituitary-adrenal axis measures (cortisol awakening response, circadian cortisol slope, cortisol levels at cognitive assessment) at each visit (baseline, week 12, and week 24).

Repeated measurements at the same time points will be obtained with a neurocognitive battery based on the CANTAB cognitive battery for schizophrenia, that includes 8 cognitive tasks: Attention Switching Task (AST; assessing attention and response latencies); One Touch Stockings of Cambridge (OTS; assessing executive functioning: spatial planning and working memory); Paired Associates Learning (PAL; assessing visual memory and new learning); Reaction Time (RTI; assessing reaction time: motor and mental response speeds, as well as measures of movement time, reaction time, response accuracy and impulsivity); Rapid Vision Information Processing (RVP; assessing sustained attention); Emotion Recognition Task (ERT; assessing theory of mind processes); Spatial Working Memory (SWM; assessing Spatial Working Memory: retention and manipulation of visuospatial information, strategy and working memory errors); Verbal Recognition Memory (VRM; assessing verbal memory and new learning). Cognitive assessment will be performed between 3 p.m. and 5 p.m. Psychopathological assessment at each visit (baseline, 12 weeks and 24 weeks) will be assessed with the Positive and Negative Syndromes Scale (PANSS) and the Calgary Depression Scale for Schizophrenia (CDSS). The social performance will be assessed at each visit with the Personal Performance Scale (PSP). Assessments will be conducted by trained personnel who will remain blind to the group assignment.

Linear mixed models will be used to explore whether hormonal or inflammatory biomarkers are associated with cognitive changes after the intervention (CRT). The model will test the fixed effects for the intervention (CRT vs TAU), time (baseline visit vs 3-month visit), and the studied hormones, as well as their interactions. Random effects will be considered for each participant. Two analyses will be conducted:

1. Primary analysis: randomized parallel phase (intention-to-treat analysis; CRT vs TAU; first 3 months).

   All participants will be included, independently of whether they completed CRT or not.
2. Secondary analysis: pre-post changes in CRT (per-protocol analysis; CRT only; 3 months).

This secondary analysis will include a subgroup of patients who have completed at least one-third of the CRT sessions. For this analysis, those patients receiving CRT in the first wave (randomized parallel phase) or second wave (after the cross-over) will be grouped.

ELIGIBILITY:
Inclusion Criteria:

* Psychotic disorder meeting Diagnostic and Statistical Manual of Mental Disorders - 4th edition (DSM-IV) criteria for any of the following diagnoses: schizophrenia, schizoaffective disorder, bipolar disorder, and psychotic disorder not otherwise specified.
* Recent-onset psychosis (< 3 years of illness).
* Outpatients with stable illness (<4 points in each positive item of the Positive and Negative Syndrome Scale [PANSS]).
* Being on community treatment for at least 4 weeks.

Exclusion Criteria:

* Refusal to participate.
* Severe neurological disease or intellectual disability.
* Pregnancy.
* Substance-induced psychosis.
* History of severe traumatic brain injury.
* Current treatment with glucocorticoids.
* Visual deficits or language difficulties that could influence cognitive assessment and intervention.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Plasma cortisol concentrations | 3 months
  Correlation between cognitive changes, assessed with the CANTAB Cognitive battery for schizophrenia, and plasma cortisol concentrations.
Cortisol awakening response | 3 months
  Correlation between cognitive changes, assessed with the CANTAB Cognitive battery for schizophrenia, and the cortisol awakening response.
Diurnal cortisol slope | 3 months
  Correlation between cognitive changes, assessed with the CANTAB Cognitive battery for schizophrenia, and the diurnal cortisol slope (calculated as the slope between salivary cortisol between awakening and 23h).
Cortisol at neuropsychological assessment | 3 months
  Correlation between cognitive changes, assessed with the CANTAB Cognitive battery for schizophrenia, and salivary cortisol at neuropsychological assessment.
Plasma prolactin concentrations | 3 months
  Correlation between cognitive changes, assessed with the CANTAB Cognitive battery for schizophrenia, and plasma prolactin concentrations.
Plasma free thyroxine (F-T4) concentrations | 3 months
  Correlation between cognitive changes, assessed with the CANTAB Cognitive battery for schizophrenia, and plasma F-T4 concentrations.
Neutrophil to lymphocyte ratio | 3 months
  Correlation between cognitive changes, assessed with the CANTAB Cognitive battery for schizophrenia, and neutrophil to lymphocyte ratio.
Plasma interleukin-6 concentrations | 3 months
  Correlation between cognitive changes, assessed with the CANTAB Cognitive battery for schizophrenia, and plasma interleukin-6 concentrations.
Plasma tumor necrosis factor alpha (TNF-alpha) concentrations | 3 months
  Correlation between cognitive changes, assessed with the CANTAB Cognitive battery for schizophrenia, and plasma TNF-alpha concentrations.

SECONDARY OUTCOMES:
Changes in plasma cortisol after a cognitive remediation therapy | 3 months
  Morning plasma cortisol concentrations will be determined. The investigators will examine longitudinal changes in plasma cortisol concentrations after a cognitive remediation therapy.
Changes in the cortisol awakening response after a cognitive remediation therapy | 3 months
  The cortisol awakening response will be measured in saliva. The investigators will examine longitudinal changes in the cortisol awakening response after a cognitive remediation therapy.
Changes in the diurnal cortisol slope after a cognitive remediation therapy | 3 months
  Salivary cortisol measures will be obtained at awakening and at 23h. The diurnal cortisol slope will be calculated between awakening and 23h. The investigators will examine longitudinal changes in the diurnal cortisol slope after a cognitive remediation therapy.
Changes in cortisol concentrations at neuropsychological assessment after a cognitive remediation therapy | 3 months
  Salivary cortisol concentrations at neuropsychological assessment will be determined. The investigators will examine longitudinal changes in cortisol concentrations at neuropsychological assessment after a cognitive remediation therapy.
Changes in plasma prolactin concentrations after a cognitive remediation therapy | 3 months
  Plasma prolactin concentrations will be determined in the morning. The investigators will examine longitudinal changes in prolactin concentrations after a cognitive remediation therapy.
Changes in plasma free thyroxine (F-T4) concentrations after a cognitive remediation therapy | 3 months
  Plasma F-T4 concentrations will be determined in the morning. The investigators will examine longitudinal changes in F-T4 concentrations after a cognitive remediation therapy.
Changes in neutrophil to lymphocyte ratio after a cognitive remediation therapy | 3 months
  Leukocyte count will be measured in plasma and the neutrophil to lymphocyte ratio will be calculated. The investigators will examine longitudinal changes in the neutrophil to lymphocyte ratio after a cognitive remediation therapy.
Changes in plasma interleukin-6 (IL-6) concentrations after a cognitive remediation therapy | 3 months
  IL-6 concentrations will be determined in plasma. The investigators will examine longitudinal changes in IL-6 concentrations after a cognitive remediation therapy.
Changes in plasma tumor necrosis factor-alpha (TNF-alpha) concentrations after a cognitive remediation therapy | 3 months
  TNF-alpha concentrations will be determined in plasma. The investigators will examine longitudinal changes in TNF-alpha concentrations after a cognitive remediation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Labad, M.D., Ph.D., Principal Investigator — Parc Taulí Hospital Universitari, Sabadell, Barcelona (Spain).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez-Gonzalo S, Turon M, Jodar M, Pousa E, Hernandez Rambla C, Garcia R, Palao D. A new computerized cognitive and social cognition training specifically designed for patients with schizophrenia/schizoaffective disorder in early stages of illness: A pilot study. Psychiatry Res. 2015 Aug 30;228(3):501-9. doi: 10.1016/j.psychres.2015.06.007. Epub 2015 Jun 18. PMID 26163731